CLINICAL TRIAL: NCT02184234
Title: A 6-week, Open, Multicentre Safety Trial to Evaluate the Tolerability Profile of Antistax® Film Coated Tablets (Extr. Vitis Viniferae Siccum), 360 mg/Day Per os, in Male and Female Patients Suffering From Chronic Venous Insufficiency
Brief Title: Tolerability of Antistax® in Patients Suffering From Chronic Venous Insufficiency (CVI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1138.5
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — Antistax

ARMS (1):
- Antistax film coated tablets (Experimental)
  Interventions: Drug: Antistax film coated tablets

INTERVENTIONS:
Drug: Antistax film coated tablets

SUMMARY:
Main objective: Safety and tolerability of Antistax® film coated tablets

Secondary objective: Effect of Antistax® film coated tablets on subjective symptoms of chronic venous insufficiency

ELIGIBILITY:
Inclusion Criteria:

* Chronic venous insufficiency stage I or II according to Widmer, e.g., resulting in lower-leg oedema
* Male or female out-patients of any ethnic origin
* Age ranging from 25 to 75 years

Exclusion Criteria:

* Known hypersensitivity to any ingredients of the study medication
* Oedema(s) of non-venous origin, e.g., due to cardiac insufficiency, lymphoedema or decompensated cardiac insufficiency, orthopaedic disturbances
* Florid venous ulcers
* Arterial occlusive disease, irrespective of the severity
* Phlebitis or thrombophlebitis
* Clinical indication for an acute phlebologic intervention, e.g., compressive treatment, phlebectomy, etc.
* Evidence of diabetic micro-angiopathy or polyneuropathy in medical history
* Poor general health (based on the investigator's judgement)
* Addiction to alcohol abuse
* Mental illness and inability (or limited ability) to work, or inability (or limited ability) to follow spoken or written explanations concerning the trial
* Women of child-bearing age not using any reliable contraceptive methods
* Pregnant or lactating women
* Patients previously enrolled in the present study or participating in another clinical study, or who had taken part in another study within the previous 90 days
* Patients receiving compression therapy, high-ceiling diuretics (e.g., furosemide), or any other anti-CVI preparations (e.g., vasoprotectives to treat varicosis, such as heparin-containing preparations, sclerosing agents, or bioflavonoids other than the study medication) during the trial. Medications or measures for CVI had to be stopped 14 day prior to intake of study medication.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2001-06; Primary Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Number and intensity of serious and non-serious Adverse Events | up to 6 weeks

SECONDARY OUTCOMES:
Global tolerability assessment by the patient and investigator | after 42 days of treatment
Vital sign parameters (blood pressure and pulse rate) | at screening and after 6 weeks
Subjective symptoms rated on a 10-cm Visual Analog Scale (VAS) | Baseline and after 6 weeks
Global assessment of efficacy by the patient and investigator | after 6 weeks